CLINICAL TRIAL: NCT06967272
Title: Evaluating the Immunogenicity and Safety of the Oral Hexavalent Reassortant Rotavirus Attenuated Live Vaccine (Vero Cells) in Healthy Infants Via a Randomized, Double-blind, Active-controlled Phase II Clinical Trial.
Brief Title: PhaseⅡClinical Trial of Oral Hexavalent Reassortant Rotavirus Attenuated Live Vaccine (Vero Cells)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-RV-2001
Record Dates: First submitted 2025-04-26; First posted 2025-05-13 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Rotavirus Gastroenteritis
Keywords: Phase II; Immunogenicity; Safety; Randomized Controlled Trial; Rotavirus gastroenteritis; Vaccine
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose (Experimental): The experimental vaccine will be administered in three doses, with a 28-day interval between each dose.
  Interventions: Biological: Oral hexavalent reassortant rotavirus attenuated live vaccine
- High dose (Experimental): The experimental vaccine will be administered in three doses, with a 28-day interval between each dose.
  Interventions: Biological: Oral hexavalent reassortant rotavirus attenuated live vaccine
- Control (Active Comparator): The controlled vaccine will be administered in three doses, with a 28-day interval between each dose.
  Interventions: Biological: Oral pentavalent reassortant rotavirus attenuated live vaccine (controlled)

INTERVENTIONS:
Biological: Oral hexavalent reassortant rotavirus attenuated live vaccine — Oral hexavalent reassortant rotavirus attenuated live vaccine (low-dose) three doses administered orally
  Arms: Low dose
Biological: Oral hexavalent reassortant rotavirus attenuated live vaccine — Oral hexavalent reassortant rotavirus attenuated live vaccine (high-dose) three doses administered orally
  Arms: High dose
Biological: Oral pentavalent reassortant rotavirus attenuated live vaccine (controlled) — The controlled vaccine three doses administered orally
  Arms: Control

SUMMARY:
The Phase II clinical trial of the oral hexavalent reassortant rotavirus attenuated live vaccine (Vero Cells) will be conducted in infants aged 6 to 12 weeks. This study will evaluate the immunogenicity and safety of the investigational vaccine in healthy infants through a randomized, double-blind, active-controlled trial.

DETAILED DESCRIPTION:
The Phase II clinical trial is a randomized, double-blind, active-controlled study conducted in healthy infants to evaluate the immunogenicity and safety of the investigational vaccine. The investigational vaccine is available in both high-dose and low-dose formulations. The control vaccine is the orally administered pentavalent reassortant rotavirus attenuated live vaccine (Vero Cells) produced by Merck Sharp & Dohme Corp.

This study plans to recruit 400 infants aged 6 to 12 weeks. All participants will be randomly assigned to the low-dose investigational group, high-dose investigational group, and active-controlled group, respectively.The immunization schedule for both the investigational vaccine and controlled vaccine consists of three doses administered at 28-day intervals.

Blood samples will be collected at predefined time points to evaluate the immunogenicity of the investigational vaccine. Adverse events (AEs) will be collected for all participants from the first vaccination until 42 days after the last dose, while serious adverse events (SAEs) and adverse events of special interest (AESIs) will be monitored for 12 months.

A safety monitoring sub-cohort will be established, with stool samples collected daily for 14 days after each vaccination to assess vaccine virus shedding, duration and patterns of viral shedding, potential reassortment and reversion to virulence of the rotavirus vaccine strains

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants aged 6 to 12 weeks.
2. The legal guardian(s) is/are capable of understanding and voluntarily signing the informed consent form.
3. The legal guardian(s) is/are willing and able to comply with all follow-up visits, sample collection, vaccination, and other study procedures.
4. Able to provide valid legal identification documents.

Exclusion Criteria:

1. Previous vaccination with any rotavirus vaccine.
2. History of rotavirus infection.
3. Gestational age <37 weeks or ≥42 weeks at birth.
4. History of dystocia, neonatal asphyxia requiring resuscitation, or neurological impairment at birth.
5. Known hypersensitivity to any vaccine component (e.g., urticaria, dyspnea, angioedema).
6. Current diarrhea, vomiting, or other gastrointestinal disorders; gastroenteritis or any acute/chronic illness exacerbation within 7 days prior to vaccination; ongoing antibiotic/antiviral therapy.
7. History of intussusception or chronic gastrointestinal diseases, including congenital malformations predisposing to intussusception (e.g., Meckel's diverticulum).
8. Congenital malformations, developmental disorders, genetic defects, severe malnutrition, malignancies, or significant chronic conditions (e.g., Down syndrome, diabetes, sickle cell anemia, neurological disorders, Guillain-Barré syndrome).
9. Autoimmune or immunodeficiency diseases (including but not limited to asplenia, functional asplenia, HIV infection).
10. Household members with immunodeficiency/immunosuppression or undergoing/scheduled for immunosuppressive/cytotoxic therapy.
11. Coagulation disorders (e.g., clotting factor deficiencies, platelet abnormalities).
12. Immunosuppressive therapy for ≥14 days post-birth (prednisone ≥2mg/kg/day or equivalent), immunomodulatory/cytotoxic therapy, or planned use during the study.
13. History of severe neurological/psychiatric disorders (e.g., epilepsy, non-febrile seizures, convulsions) or relevant family history.
14. Postnatal administration of immunoglobulins/blood products (except hepatitis B immunoglobulin) or planned use during the study.
15. Previous participation in other investigational drug/vaccine studies or planned use during this study.
16. Receipt of live-attenuated vaccines within 14 days or subunit/inactivated vaccines within 7 days prior to enrollment.
17. Axillary temperature ≥38.0°C within the past 3 days.
18. Fever on scheduled vaccination day (axillary temperature >37.0°C; measured ≥30 minutes post-feeding).
19. Currently or planning to participate in other vaccine or drug clinical trials.
20. Any other factors that the investigator deems unsuitable for participation in the clinical trial.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the immunogenicity of the investigational vaccine at different doses | 28 days after the full vaccination course
  The seroconversion rate of IgA antibodies against vaccine-type rotavirus in serum
Evaluate the safety of the investigational vaccine at different dose | 0 day after the first dose till 42 days after the last dose
  Incidence of adverse events/reactions

SECONDARY OUTCOMES:
Evaluate the immunogenicity of the investigational vaccine at different doses | 28 days after the full vaccination course
  The positivity rate of serum anti-vaccine-type rotavirus IgA antibodies
Evaluate the immunogenicity of the investigational vaccine at different doses | 28 days after the full vaccination course
  The geometric mean concentration (GMC) of serum anti-vaccine-type rotavirus IgA antibodies
Evaluate the immunogenicity of the investigational vaccine at different doses | 28 days after the full vaccination course
  The geometric mean increase (GMI) of serum anti-vaccine-type rotavirus IgA antibodies
Evaluate the immunogenicity persistence of the investigational vaccine at different doses | 12 months after the full vaccination course
  The geometric mean concentration (GMC) of serum anti-vaccine-type rotavirus IgA antibodies
Evaluate the immunogenicity persistence of the investigational vaccine at different doses | 12 months after the full vaccination course
  The positivity rate of serum anti-vaccine-type rotavirus IgA antibodies
Evaluate the safety of the investigational vaccine at different dose | 0-30 minutes after each dose
  Incidence of adverse events/reactions
Evaluate the safety of the investigational vaccine at different dose | 0-14 days after each dose
  Incidence of adverse events/reactions
Evaluate the safety of the investigational vaccine at different dose | The first dose to 12 months after full vaccination
  Incidence of serious adverse events (SAEs) and adverse events of special interest (AESIs)
Evaluate the fecal shedding of investigated vaccine strain after vaccination | 0-14 days after each dose
  The shedding rate of the rotavirus vaccine strain in the stool.
Evaluate the fecal shedding of investigated vaccine strain after vaccination | 0-14 days after each dose
  The shedding duration of the rotavirus vaccine strain in the stool.
Evaluate the reassortment and reversion of the rotavirus vaccine strain in stool samples after vaccination | 0-14 days after each dose
  The incidence of reassortment and reversion of the rotavirus vaccine strain in stool samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei Provincial Center for Disease Control and Prevention, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided